CLINICAL TRIAL: NCT01328808
Title: Metabolism and Toxicity of Acetaminophen in Preterm Infants
Brief Title: Metabolism and Toxicity of Acetaminophen
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: John van den Anker (Other)
Responsible Party: Sponsor-Investigator, John van den Anker, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4839 - APAP
Record Dates: First submitted 2011-03-30; First posted 2011-04-05 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2021-12

CONDITIONS: Pain
Keywords: Acetaminophen; Preterm Infants
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- group 2 Pain management (Experimental): In preterm and term neonates with a GA of 28 weeks or more a 15 mg/kg dose of APAP will be given every 8 hrs by an intravenous infusion over 30-minute.
  In preterm and term neonates with a GA of less than 28 weeks 15 mg/kg dose of APAP will be given every 12 hrs by an intravenous infusion over 30-minute
  Interventions: Drug: Acetaminophen/APAP

INTERVENTIONS:
Drug: Acetaminophen/APAP — In preterm and term neonates with a GA of 28 weeks or more a 15 mg/kg dose of APAP will be given every 8 hrs by an intravenous infusion over 30-minute.
  In preterm and term neonates with a GA of less than 28 weeks a 15 mg/kg dose of APAP will be given every 8 hrs by an intravenous infusion over 30-minute
  Other Names: Tylenol

SUMMARY:
The purpose of this study is to investigate how acetaminophen (APAP) is released into the urine and blood; to determine how the blood levels of acetaminophen and its breakdown products affect the preterm infant's health; to decrease adverse drug reactions; and to collect data on how the genetic make-up or characteristics affect how APAP is handled within the preterm infant. By taking several blood and urine samples during the study, we will be able to check the blood levels (called pharmacokinetics) of APAP in preterm babies.

DETAILED DESCRIPTION:
Study procedures: The decision to replace standard intravenous morphine therapy with APAP will be made by the attending neonatologist.

Length of participation: 60 hours. No patient will be prescribed the medication specifically for the study purposes in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Preterm and term neonates of both genders and all races
* a postnatal age of less than 28 days
* GA's of from 22 to less than 37 weeks
* an indwelling (peripheral or umbilical) arterial line
* a clinical indication for intravenous administration of pain relief medication

Exclusion Criteria:

* Neonates with severe asphyxia
* grade III or IV intraventricular hemorrhage, major congenital malformations/facial malformations (e.g., cleft lip and palate),
* neurological disorders
* those receiving continuous or intermittent neuromuscular blockers
* clinical or biochemical evidence of hepatic renal failure (including systemic hypoperfusion)

Ages: 22 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
primary endpoint PK analysis | 48 hours
  Blood and urine levels of APAP and metabolites

SECONDARY OUTCOMES:
Developmental stage | 48 hours
  To assess both the magnitude and statistical significance of any evidence of relationship between developmental stage and toxicity-associated metabolite levels.
  The analyses will also hold constant APAP dose, BID or TID and possible confounding variables such as birth order, maternal smoking status, and maternal age. We will plot the relationship between stage of development and measures of APAP Metabolism, taken at different gestational and postnatal ages. A hierarchical, cross sectional time series models will be used.

CONTACTS AND LOCATIONS:
Overall Officials: John N van den Anker, MD, PhD, Principal Investigator — Children's National Research Institute
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Childrens Research Institute, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Yes
There is no plan to share individual participant data. Preliminary data published Published manuscripts in 2015 & 2016

REFERENCES:
- [Result] Cook SF, Stockmann C, Samiee-Zafarghandy S, King AD, Deutsch N, Williams EF, Wilkins DG, Sherwin CM, van den Anker JN. Neonatal Maturation of Paracetamol (Acetaminophen) Glucuronidation, Sulfation, and Oxidation Based on a Parent-Metabolite Population Pharmacokinetic Model. Clin Pharmacokinet. 2016 Nov;55(11):1395-1411. doi: 10.1007/s40262-016-0408-1. PMID 27209292
- [Result] Cook SF, King AD, van den Anker JN, Wilkins DG. Simultaneous quantification of acetaminophen and five acetaminophen metabolites in human plasma and urine by high-performance liquid chromatography-electrospray ionization-tandem mass spectrometry: Method validation and application to a neonatal pharmacokinetic study. J Chromatogr B Analyt Technol Biomed Life Sci. 2015 Dec 15;1007:30-42. doi: 10.1016/j.jchromb.2015.10.013. Epub 2015 Oct 31. PMID 26571452
- [Result] Cook SF, Roberts JK, Samiee-Zafarghandy S, Stockmann C, King AD, Deutsch N, Williams EF, Allegaert K, Wilkins DG, Sherwin CM, van den Anker JN. Population Pharmacokinetics of Intravenous Paracetamol (Acetaminophen) in Preterm and Term Neonates: Model Development and External Evaluation. Clin Pharmacokinet. 2016 Jan;55(1):107-19. doi: 10.1007/s40262-015-0301-3. PMID 26201306